CLINICAL TRIAL: NCT01311908
Title: Effect of a Roux-en-Y Reconstruction on Reflux Esophagitis After Pancreaticoduodenectomy
Brief Title: Incidence of Reflux Esophagitis After Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tien Yu-Wen, M.D., Ph.D., National Taiwan University Hospital
Other Study IDs: 201005058R
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Reflux Esophagitis
Keywords: Pancreaticoduodenectomy; Roux-en-Y reconstruction; Reflux esophagitis
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — esophageal mucosal biopsy for Real-Time PCR for COX-2 activity
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery, Roux-en-Y , reflux esophagitis: Patients with roux-en-Y reconstruction (study group)
  Interventions: Procedure: Methods of gastrojejunostomy reconstruction
- surgery, traditional gastrojejunostomy: Traditional gastrojejunostomy reconstruction (control group).

INTERVENTIONS:
Procedure: Methods of gastrojejunostomy reconstruction — Roux-en-Y reconstruction in pancreaticoduodenectomy
  Other Names: Reconstruction of gastrojejunostomy; Roux-en-Y anastomosis versus gastrojejunostomy only
  Groups: Surgery, Roux-en-Y , reflux esophagitis

SUMMARY:
Reflux esophagitis is a common complication following distal gastrectomy. According to the investigators preliminary data, an Roux-en--Y gastrointestinal reconstruction in pancreaticoduodenectomy is associated with higher rates of reflux esophagitis. In this study, the investigators will investigate the incidence of reflux esophagitis after above procedure by the 24-h pH monitoring of esophagogastric junction.

DETAILED DESCRIPTION:
Reflux esophagitis is a common complication following distal gastrectomy. Recently, an Roux-en--Y gastrointestinal reconstruction has been used increasingly to prevent reflux esophagitis; however, reflux esophagitis after pancreaticoduodenectomy (also including distal gastrectomy) has never been studied.

In our preliminary retrospective study of 371 patients having PD (158 standard PD and 213 pylorus-preserving PD) at our hospital, after a median follow-up of 20 months (range, 2-110 months), 40 patients (10.8%) developed reflux esophagitis - 15 (9.5%) in the standard PD group, and 25 (11.7%) in the PPPD group. Multivariate logistic regression analysis revealed the only significant factors related to reflux esophagitis is Roux-en-Y gastrointestinal reconstruction independent of preservation of the pylorus.

To our surprise, there is no significant difference in occurrence of GERD between patients after standard PD (15 of 158 patient) and PPPD (25 of 313 patients, P=0.49). We postulate reflux esophagitis following a PPPD in patients without past history of GERD is most likely caused by disruption of reflux-preventing systems at the gastroesophageal junction, thereby allowing reflux of gastric acid into esophagus. If the postulation is true, GERD after PPPD should be acidic in nature. To test this hypothesis we propose a prospective randomized study to compare preoperative and postoperative parameters, including esophageal morphology, bile acid concentration, trypsin activity of esophageal refluxate, COX2 mRNA expression of lower esophageal mucosa, and 24 hour pH monitor of lower esophagus.

Moreover, to test the effect of a Roux-en-Y reconstruction to prevent GERD after PD, studied patients will be randomized into Roux-en-Y and control groups to study inter-group differences in incidence of GERD and marginal ulcer after PD.

Acidic GERD should be treated with proton pump inhibitor. In contrast, alkaline GERD should be treated with pro-kinetic agent such as primperan and mopride. With this study, we can learn more about the nature of post-PD GERD following various gastrointestinal reconstructions and can give patient more personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years and planned PD for a lesion of either the pancreatic head or the periampullary region

Exclusion Criteria:

* history of abdominal or pelvic radiation
* hepatic dysfunction (Child-Pugh > 2)
* renal dysfunction (serum creatinine concentration > 3 mg/L, hemodialysis, or both)
* cardiac dysfunction (New York Heart Association functional class > III, stroke history)
* pregnancy
* history of intestinal anastomosis of the large bowel without a diverting stoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tudy the effect of a Roux-en-Y reconstruction on GERD and marginal ulcer after pancreaticoduodenectomy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of reflux esophagitis | 3 months
  Use panendiscopy to assess the reflux esopagitis

SECONDARY OUTCOMES:
Incidenc of marginal ulcer | 3 months
  Use endoscopy to assess the marginal ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wen Tien, M.D., Ph.D., Principal Investigator — Department of surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan